CLINICAL TRIAL: NCT01665612
Title: The Evaluation of the Clinical and Subjective Performance of Three Different Contact Lens Care Solutions With Silicon Hydrogel Lenses
Brief Title: The Clinical and Subjective Performance of Three Different MPDS With Silicon Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnsusp Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: FI-2012
Record Dates: First submitted 2012-08-08; First posted 2012-08-15 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Adverse Reaction to Contact Lens Solution
Keywords: Contact lens; Care solution; MPDS; comfort

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MPDS1 (Experimental): Contact lens care solution
  Interventions: Device: Contact lens care solution
- MPDS2 (Active Comparator): Contact lens care solution
  Interventions: Device: Contact lens care solution
- MPDS3 (Active Comparator): Contact lens care solution
  Interventions: Device: Contact lens care solution

INTERVENTIONS:
Device: Contact lens care solution — Comparison of clinical and subjective performation of the contact lens care solutions used with two types of contact lenses

SUMMARY:
The purpose of the clinical investigation is to assess the clinical and subjective performance of three novel multipurpose disinfecting solutions (MPDS) in daily wear with two silicone hydrogel contact lenses (Lotrafilcon B and Comfilcon A).

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* experienced contact lens user
* good health (self-reported)

Exclusion Criteria:

* eye disease or eye operations
* pregnancy
* medication that can affect sight

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance | 1 month
  TBUT, conjunctival and limbal hyperemia, corneal vascularization, epithelial and stromal oedema, corneal infiltrates, endothelial regularity, corneal staining and papillar conjunctivitis

SECONDARY OUTCOMES:
Subjective performance | 1 month
  E.g. Comfort

CONTACTS AND LOCATIONS:
Overall Officials: Riikka Järvinen, PhD, Study Director — University of Turku, Finland; Finnsusp Ltd, Finland; Hanna Vaahtoranta-Lehtonen, Dr. Ophth., Principal Investigator — Turku University Hospital
Locations (1):
- Raision Näkökulma, Raisio, Finland